CLINICAL TRIAL: NCT03146962
Title: A Phase II Study of High Dose Vitamin C Intravenous Infusion in Patients With Resectable or Metastatic Solid Tumor Malignancies
Brief Title: High Dose Vitamin C Intravenous Infusion in Patients With Resectable or Metastatic Solid Tumor Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1610017688
Record Dates: First submitted 2017-04-27; First posted 2017-05-10 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort A: Vitamin C + Surgery (Experimental): Vitamin C infusion will be administered intravenously at 1.25 g/kg for 4 days per week for 2-4 consecutive weeks.
  Interventions: Drug: Vitamin C
- Cohort B: Vitamin C Only (Experimental): Vitamin C infusion will be administered intravenously at 1.25 g/kg for 4 days per week for up to 6 months.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 1 (Experimental): Vitamin C will be administered at a dose of 0.5 g/kg intravenously for 4 days /week for 1-2 weeks prior to and following Y90 therapy for a total of 4 weeks of vitamin C.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 2 (Experimental): Vitamin C will be administered at a dose of 0.75 g/kg intravenously for 4 days /week for 1-2 weeks prior to and following Y90 therapy for a total of 4 weeks of vitamin C.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 3 (Experimental): Vitamin C will be administered at a dose of 0.75 g/kg intravenously for 4 days /week for 1-2 weeks prior to and following Y90 therapy for a total of 4 weeks of vitamin C. A single dose of Vitamin C at 0.5g/kg will also be administered on the day of Y90 radioembolization, administered prior to or within 24 hours of a Y90 treatment.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 4 (Experimental): Vitamin C will be administered at a dose of 1 g/kg intravenously for 4 days /week for 1-2 weeks prior to and following Y90 therapy for a total of 4 weeks of vitamin C. A single dose of Vitamin C at 0.5g/kg will also be administered on the day of Y90 radioembolization, administered prior to or within 24 hours of a Y90 treatment.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 5 (Experimental): A single dose of Vitamin C at 0.75g/kg will be administered on the day of Y90 radioembolization, administered prior to or within 24 hours of a Y90 treatment. Vitamin C will also be administered at a dose of 1 g/kg intravenously for 4 days/week for 1-2 weeks following Y90 therapy.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 6 (Experimental): A single dose of Vitamin C at 0.75g/kg will be administered on the day of Y90 radioembolization, administered prior to or within 24 hours of a Y90 treatment. Vitamin C will also be administered at a dose of 1.25 g/kg intravenously for 4 days/week for 1-2 weeks following Y90 therapy.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 7 (Experimental): A single dose of Vitamin C at 1g/kg will be administered on the day of Y90 radioembolization, administered prior to or within 24 hours of a Y90 treatment. Vitamin C will also be administered at a dose of 1.25 g/kg intravenously for 4 days/week for 1-2 weeks following Y90 therapy.
  Interventions: Drug: Vitamin C
- Cohort C: Vitamin C + Y-90 Dose Level 8 (Experimental): A single dose of Vitamin C at 1.25g/kg will be administered on the day of Y90 radioembolization, administered prior to or within 24 hours of a Y90 treatment. Vitamin C will also be administered at a dose of 1.25 g/kg intravenously for 4 days/week for 1-2 weeks following Y90 therapy.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Vitamin C infusion will be administered intravenously at 1.25 g/kg for 4 days per week for 2-4 consecutive weeks (cohort A) or up to 6 months (cohort B). Cohort C will receive high dose vitamin C for 1-3 weeks. During week 1 vitamin C infusion and Y90 radioembolization of hepatic metastases will occur same day.
  Other Names: Ascorbic Acid

SUMMARY:
This is a multicenter, single arm, 3-cohort, open-label trial of high dose Vitamin C intravenous infusion in subjects with solid tumor malignancies who are eligible for resection (cohort A) or with extended RAS (e.g.KRAS or NRAS) or BRAF mutation metastatic cancer who have received prior systemic treatment (cohort B). Cohort C will involve patients with colorectal cancer having an extended RAS or BRAF mutation who are amenable for localregional therapy of hepatic metastases with Yttrium-90 radioembolization.

DETAILED DESCRIPTION:
This clinical trial is for men and women with resectable or metastatic solid tumor malignancies. The objective of the study is to investigate whether high dose vitamin C infusion leads to pathological tumor response in resectable colorectal, pancreatic, and lung cancer (cohort A) or objective tumor response in KRAS or BRAF mutant solid tumors (cohort B). For Cohort C, the primary objective is to determine that maximal tolerated dose of the combination of high dose vitamin C with Y90 radioembolization for patients solid tumor malignancies and liver metastases amenable to local-regional therapy

Patients in cohort A receive a high dose vitamin C infusion for 4 days per week for 2-4 consecutive weeks prior to surgery. Patients in cohort B receive high dose vitamin C infusion for 4 days per week for up to 6 months or disease progression. Cohort C will receive high dose vitamin C for 1-3 weeks. During week 1 vitamin C infusion and Y90 radioembolization of hepatic metastases will occur same day.

A tumor sample will be resected after completion of study drug (high dose vitamin C infusion) treatment to examine the effects of study drug (Cohort A only). In addition, organoids will be grown in vitro and continue to be treated with vitamin C added in culture medium to examine tumor response. The resected tumor in this study will

Key eligibility:

* Men and women age 18 and older
* Patients with histologically proven early stage or locally advanced colorectal adenocarcinoma, lung cancer or pancreatic cancer, who are eligible for resection, and have not received chemotherapy or radiotherapy (cohort A) Patients with inoperable, metastatic, KRAS or BRAF mutant colorectal adenocarcinoma, lung cancer and pancreatic cancer, who have received at least 1 line of treatment for metastatic disease (cohort B)
* Patients with metastatic cancer with an extended RAS (e.g. KRAS or NRAS) or BRAF mutation with liver metastases amenable to Y90 radioembolization (cohort C).

ELIGIBILITY:
Inclusion Criteria

* Male or female ≥ 18 years of age.
* Patients with histologically proven early stage or locally advanced colorectal adenocarcinoma, lung cancer or pancreatic cancer, who are eligible for resection (cohort A).
* Patients with inoperable, metastatic extended RAS (e.g. KRAS or NRAS) or BRAF mutant colorectal adenocarcinoma, lung cancer and pancreatic cancer, or other solid tumor, who have received at least 1 line of treatment for metastatic disease (cohort B).
* Patients with metastatic cancer with an extended RAS (e.g. KRAS or NRAS) or BRAF mutation with liver metastases amenable to Y90 radioembolization (cohort C).
* ECOG performance status 0-1.
* Life expectancy of at least 6 months.
* All women of child-bearing potential and all sexually active male patients must agree to use effective contraception.

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure (NYHA class III and IV), uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements (Appendix B: New York Heart Association (NYHA) Classifications).
* Patients with active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, unstable angina pectoris, or uncontrolled congestive heart failure (NYHA class III and IV) (Appendix B: New York Heart Association (NYHA) Classifications).
* Patients who have received an investigational drug within 21 days of the first dose of study drug.
* Patients who are pregnant or lactating.
* Patients who are known to be positive for the human immunodeficiency virus (HIV). The effect of Vitamin C on HIV medications is unknown. Note: HIV testing is not required for eligibility, but if performed previously and was positive, the patient is ineligible for the study.
* Patient who are receiving drugs which are known to interact with Vitamin C, potential risk and eligibility will be evaluated individually by the investigator. a. Most of the known interactions with vitamin C are from oral use and acidification of the stomach lining. There are few known interactions with high dose intravenous vitamin C. We recommend not using deferoxamine as there may be an association with ventricular dysfunction (unknown mechanism).
* Patients who have uncontrolled or severe hyponatremia, hypernatremia, SIADH, hypokalemia, hyperkalemia, hypomagnesemia, or hypermagnesemia
* Patients who have uncontrolled or severe coagulopathies or a history of clinically significant bleeding within the past 6 months, such as hemoptysis, epistaxis, hematochezia, hematuria, or gastrointestinal bleeding.
* Patients who require therapeutic doses of warfarin
* Patients who have uncontrolled seizure disorder, ascites, iron overload, edema, or dehydration.
* Patients who have glucose-6-phosphate dehydrogenase (G6PD) deficiency, hereditary spherocytosis, or other conditions predisposing patient to hemolysis.
* Patients who have a known history of recurrent oxalate renal calculi or multiple oxalate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: Vitamin C + Surgery | Cohort B: Vitamin C Only | Cohort C: Vitamin C + Y-90 Dose Level 1 | Cohort C: Vitamin C + Y-90 Dose Level 2 | Cohort C: Vitamin C + Y-90 Dose Level 3 | Cohort C: Vitamin C + Y-90 Dose Level 4 | Cohort C: Vitamin C + Y-90 Dose Level 5 | Cohort C: Vitamin C + Y-90 Dose Level 6 | Cohort C: Vitamin C + Y-90 Dose Level 7 | Cohort C: Vitamin C + Y-90 Dose Level 8
Started | 7 | 21 | 3 | 3 | 4 | 3 | 3 | 7 | 3 | 7
Completed | 5 | 15 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 6
Not Completed | 2 | 6 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID Precautions | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Started New Treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Vitamin C + Surgery | Cohort B: Vitamin C Only | Cohort C: Vitamin C + Y-90 Dose Level 1 | Cohort C: Vitamin C + Y-90 Dose Level 2 | Cohort C: Vitamin C + Y-90 Dose Level 3 | Cohort C: Vitamin C + Y-90 Dose Level 4 | Cohort C: Vitamin C + Y-90 Dose Level 5 | Cohort C: Vitamin C + Y-90 Dose Level 6 | Cohort C: Vitamin C + Y-90 Dose Level 7 | Cohort C: Vitamin C + Y-90 Dose Level 8 | Total
Number analyzed (Participants) | 7 | 21 | 3 | 3 | 4 | 3 | 3 | 7 | 3 | 7 | 61
Age, Continuous [Median (Full Range); unit: years] | 49.02 [44.09 to 77.89] | 60.72 [40.98 to 87.84] | 54.51 [48.49 to 71.18] | 55.5 [42.51 to 71.66] | 75.66 [69.04 to 77.85] | 48.46 [46.86 to 65.21] | 77.73 [68.09 to 79.43] | 58.05 [43.96 to 70.74] | 69.92 [66.11 to 69.92] | 58.94 [50.15 to 74.46] | 61.66 [40.98 to 87.84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 1 | 1 | 2 | 0 | 2 | 3 | 1 | 2 | 31
  Male | 2 | 7 | 2 | 2 | 2 | 3 | 1 | 4 | 2 | 5 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 10
  Not Hispanic or Latino | 6 | 16 | 3 | 2 | 2 | 2 | 3 | 7 | 2 | 7 | 50
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 6
  White | 5 | 14 | 3 | 2 | 2 | 3 | 3 | 5 | 2 | 5 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Region of Enrollment [Number; unit: participants]
  United States | 7 | 21 | 3 | 3 | 4 | 3 | 3 | 7 | 3 | 7 | 61

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response Based on Tumor Regression Grading in Cohort A Patients
Description: Number of patients with partial or complete pathological response in surgically resected tumor tissue: Pathological response rate is the number of patients with partial or complete pathological response in surgically resected tumor tissue. Pathologic response was assessed by tumor regression grade. This is a pathologic assessment of the amount of residual cancer cells in the specimen and the degree of fibrosis in the sample specimen. A completer response is 0% residual cancer cells. A partial response is 10-50% residual cancer cells, and no response is >50% residual cancer cells within the tumor specimen.
Time Frame: cohort A - 8 weeks
Population: Only the 6 patients who had surgery from Cohort A, and thus had evaluable tissue, were analyzed for this measure. Participants in Cohort B and C did not undergo surgery, and were thus not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Vitamin C + Surgery
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: 3-month Disease Control Rate (DCR) Will be Evaluated Using RECIST v 1.1 in Cohort B Patients.
Description: Percentage of patients with complete response, partial response, or stable disease as a result of their therapy at 3 months
Time Frame: Cohort B - 3 months
Population: DCR was not collected for Cohort A or Cohort C. 5 participants from Cohort B were missing scans and were therefor unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B: Vitamin C Only
Number analyzed (Participants) | 16
Participants | 1

3. Primary Outcome: Maximal Tolerated Dose of High Dose Vitamin C in Combination With Y90 Radioembolization
Description: Maximal tolerated dose will be evaluated by assessment of dose limiting toxicities for multiple dose levels. Dose limiting toxicity will be defined as any grade 3-4 adverse event possibly, probably, or definitely attributed to vitamin C therapy in the 21 days of protocol therapy. In any group of 3 patients, if one patient experiences dose limiting toxicity, the group will be expanded by 3 additional patients (eg. 6 for that group). If, at any dose level, 2 or more patients experience a dose limiting toxicity, the maximal tolerated dose will be reached, and further dose escalation will not be pursued. The dose level may then be expanded up to 10 additional patients to confirm the safety and toxicity at that dose level.
Time Frame: Cohort C - 16 weeks
Population: Only patients that received a dose of Vitamin C in Cohort C were considered evaluable. In Cohort C, 30 out of 32 participants who received vitamin C were evaluated across dose levels. Cohort A and B were not dose escalations, and therefore were not evaluated for maximum tolerated dose.
Measure: Number; unit: g/kg
Groups:
- Cohort C: Vitamin C + Y-90 (All Dose Levels): Vitamin C infusion will be administered intravenously at for 4 days per week for 1-4 weeks. Vitamin C will also be administered the same day as, or within 24 hours prior to, Y90 radioembolization of hepatic metastases.
  Vitamin C: Vitamin C infusion will be administered intravenously at 1.25 g/kg for 4 days per week for 2-4 consecutive weeks (cohort A) or up to 6 months (cohort B). Cohort C will receive high dose vitamin C for 1-3 weeks. During week 1 vitamin C infusion and Y90 radioembolization of hepatic metastases will occur same day.
Arm/Group | Cohort C: Vitamin C + Y-90 (All Dose Levels)
Number analyzed (Participants) | 30
g/kg
  Vitamin C Weekly Infusion Dose | 1.25
  Vitamin C Infusion Dose the Day of Y-90 Radioembolization | 1.25

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from registration to cancer progression or death due to any cause for up to 6 months. Cancer progression is defined using the Response Evaluation Criteria in Solid Tumors v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in non-target lesions, or the appearance of new lesions.
Time Frame: cohort B - up to 6 months
Population: Participants from Cohort A and Cohort C were not assessed for PFS. 5 participants were missing scans from Cohort B and were therefore unevaluable.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort B: Vitamin C Only
Number analyzed (Participants) | 16
days | 36 [14 to 151]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Number of patients with a partial response or complete response based on RECIST 1.1 Criteria.
Time Frame: cohort B - up to 6 months cohort C - 16 weeks
Population: For Cohort B, only 16/21 participants had complete sets of imaging scans and were therefore evaluable. Participants in Cohort A were not evaluated for ORR. In Cohort C Dose Level 3, one patient withdrew from the study early and therefore was unevaluable. For cohort C dose level 6, three patients did not have complete imaging to be evaluable. For Cohort C Dose Level one participant withdrew prior to treatment and one participant was missing scans, therefore they were not unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B: Vitamin C Only | Cohort C: Vitamin C + Y-90 Dose Level 1 | Cohort C: Vitamin C + Y-90 Dose Level 2 | Cohort C: Vitamin C + Y-90 Dose Level 3 | Cohort C: Vitamin C + Y-90 Dose Level 4 | Cohort C: Vitamin C + Y-90 Dose Level 5 | Cohort C: Vitamin C + Y-90 Dose Level 6 | Cohort C: Vitamin C + Y-90 Dose Level 7 | Cohort C: Vitamin C + Y-90 Dose Level 8
Number analyzed (Participants) | 16 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

6. Secondary Outcome: Time to Maximum Concentration and Half-life of Vitamin C (t1/2) in Hours in Cohort B
Description: The serum concentration of vitamin C was serially measured following vitamin C infusion at 1.25 g/kg at various timepoints up to 24 hours post infusion to determine the Tmax and t(1/2) in hours
Time Frame: Up to 24 hours post-infusion
Population: Pharmacokinetics data was not assessed for Cohort A or Cohort C. PK samples for 5 participants from Cohort B were not obtained and therefore only 16/21 participants were evaluable.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort B: Vitamin C Only
Number analyzed (Participants) | 16
hours
  T(max) | 2.28 (0.38)
  t(1/2) | 6.46 (1.44)

7. Secondary Outcome: Safety of High Dose Vitamin C Administration Using CTCAE 4.03.
Description: The number of participants per cohort who experienced a Grade 3 or 4 adverse event (as defined by CTCAE v4.03) that was deemed possibly, probably, or definitely related to Vitamin C.
Time Frame: Adverse events were assessed from the start of study treatment to 30 days after the last infusion of vitamin C. For Cohort A and C, this was approximately 2 months. For Cohort B this was about a 6 month duration.
Population: Overall number of participants analyzed includes any participants that were enrolled in the study and received at least one dose of Vitamin C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Vitamin C + Surgery | Cohort B: Vitamin C Only | Cohort C: Vitamin C + Y-90 Dose Level 1 | Cohort C: Vitamin C + Y-90 Dose Level 2 | Cohort C: Vitamin C + Y-90 Dose Level 3 | Cohort C: Vitamin C + Y-90 Dose Level 4 | Cohort C: Vitamin C + Y-90 Dose Level 5 | Cohort C: Vitamin C + Y-90 Dose Level 6 | Cohort C: Vitamin C + Y-90 Dose Level 7 | Cohort C: Vitamin C + Y-90 Dose Level 8
Number analyzed (Participants) | 7 | 19 | 3 | 3 | 4 | 3 | 3 | 7 | 3 | 6
Participants
  Alkaline Phosphatase Increase | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Aspartate Aminotransferase Increase | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
  Alanine Aminotransferase Increase | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Anemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hypokalemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood Bilirubin Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypertension | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Generalized Muscle Weakness | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Confusion | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Scrotal Pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Syncope | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemolysis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Concentration of Vitamin C in Hours in Cohort B
Description: The serum concentration of vitamin C was serially measured following vitamin C infusion at 1.25 g/kg at various timepoints up to 24 hours post infusion to determine the maximum concentration (Cmax) in mM.
Time Frame: Up to 24 hours post-infusion
Population: Pharmacokinetics were not assessed for Cohort A and C. PK samples for 5 participants from Cohort B were not obtained and therefore only 16/21 participants were evaluable.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Cohort B: Vitamin C Only
Number analyzed (Participants) | 16
mM | 41.19 (10.89)

9. Other Pre Specified Outcome: In Vitro Activity of Vitamin C in Tumor Organoids
Description: Molecular signature of vitamin C efficacy will be determined using RNA sequencing and compared between KRAS or BRAF mutant vs wild type tumors. Organoids will be prepared from resected tumor samples and treated with vitamin C.
Time Frame: cohort A - 8 weeks, cohort B - up to 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory Biomarker Samples From Tumor Tissue Will be Collected at the Time Points Specified in the Protocol
Description: To explore potential correlation of gene expression pattern with anti-tumor activity of vitamin C, we plan to perform RNA sequencing using surgical sample in cohort A patients who will receive vitamin C infusion pre-operatively.
Time Frame: cohort A - 8 weeks, cohort B - up to 6 months, Cohort C - 16 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Pharmacodynamic Samples From Tumor Tissue Will be Collected at the Time Points Specified in the Protocol.
Description: Immunohistochemical (IHC) staining for GLUT1 protein expression will be performed on Formalin Fixed Paraffin Embedded (FFPE) tumor tissues. Immunohistochemical (IHC) staining for phosphor-AMPK will be performed on Formalin Fixed Paraffin Embedded (FFPE) tumor tissues to assess AMPK activation.
Time Frame: cohort A - 8 weeks, cohort B - up to 6 months, Cohort C - 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the start of study treatment to 30 days after the last infusion of vitamin C. For Cohort A and C, this was approximately 2 months. For Cohort B this was about a 6 month duration. Some study participants were enrolled in the trial, but did not receive study treatment, so they are not included in the at risk population.
Description: All enrolled participants were assessed for death. Only participants treated were assessed for adverse events. Two participants that were enrolled in Cohort B Vitamin C Only were withdrawn prior to receiving study treatment. One participant that was enrolled in Vitamin C + Y-90: Dose Level 8 was withdrawn from the study before receiving study treatment. Therefore they were not included in the at risk population for adverse events, only mortality.
Groups:
- Cohort B Vitamin C Only: Vitamin C infusion will be administered intravenously at 1.25 g/kg for 4 days per week for up to 6 months.
  Vitamin C: Vitamin C infusion will be administered intravenously at 1.25 g/kg for 4 days per week for 2-4 consecutive weeks (cohort A) or up to 6 months (cohort B). Cohort C will receive high dose vitamin C for 1-3 weeks. During week 1 vitamin C infusion and Y90 radioembolization of hepatic metastases will occur same day.
Arm/Group | Cohort A: Vitamin C + Surgery | Cohort B Vitamin C Only | Cohort C: Vitamin C + Y-90 Dose Level 1 | Cohort C: Vitamin C + Y-90 Dose Level 2 | Cohort C: Vitamin C + Y-90 Dose Level 3 | Cohort C: Vitamin C + Y-90 Dose Level 4 | Cohort C: Vitamin C + Y-90 Dose Level 5 | Cohort C: Vitamin C + Y-90 Dose Level 6 | Cohort C: Vitamin C + Y-90 Dose Level 7 | Cohort C: Vitamin C + Y-90 Dose Level 8
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/21 | 0/3 | 0/3 | 0/4 | 0/3 | 0/3 | 2/7 | 0/3 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 4/19 | 0/3 | 0/3 | 0/4 | 0/3 | 0/3 | 4/7 | 0/3 | 2/6
Other Adverse Events (participants affected / at risk) | 6/7 | 18/19 | 3/3 | 3/3 | 3/4 | 3/3 | 3/3 | 7/7 | 2/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Vitamin C + Surgery (N=7) | Cohort B Vitamin C Only (N=19) | Cohort C: Vitamin C + Y-90 Dose Level 1 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 2 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 3 (N=4) | Cohort C: Vitamin C + Y-90 Dose Level 4 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 5 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 6 (N=7) | Cohort C: Vitamin C + Y-90 Dose Level 7 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 8 (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Infection (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Vitamin C + Surgery (N=7) | Cohort B Vitamin C Only (N=19) | Cohort C: Vitamin C + Y-90 Dose Level 1 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 2 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 3 (N=4) | Cohort C: Vitamin C + Y-90 Dose Level 4 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 5 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 6 (N=7) | Cohort C: Vitamin C + Y-90 Dose Level 7 (N=3) | Cohort C: Vitamin C + Y-90 Dose Level 8 (N=6)
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 2 | 2 | 1 | 2 | 2 | 4 | 0 | 1
Fatigue (General disorders) | 2 | 6 | 1 | 0 | 1 | 2 | 2 | 4 | 1 | 2
Alkaline phosphatase increased (Investigations) | 2 | 5 | 2 | 0 | 1 | 0 | 2 | 5 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 7 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2
Hypokalemia (Investigations) | 0 | 4 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 7 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 0 | 2 | 1 | 2 | 0 | 2 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Fever (General disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 3 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Edema Limbs (General disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders Other, Bleeding Gums (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Other: Cold Intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: COVID-19 Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flu Like Symptoms (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Increased Lactate Dehydrogenase (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Other: Blood in Stool (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Neuropathy, Type Unspecified (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Other: Activity Change (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Bleeding Gums (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Other: Chest Pain, unspecified (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Other: Diaphoresis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Other: Dry Heaves (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Edema face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Other: "Feeling Shaky" (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight Loss (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Chest tightness/discomfort (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Other: Tachycardia, unspecified (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Other: Loss of Hand Movement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Rash (Unspecified) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight gain (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Other: Night Sweats (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Other: Increased Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Appetite Change (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Other: Jaundice (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other: Ketosis (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03146962/Prot_SAP_000.pdf